CLINICAL TRIAL: NCT04221672
Title: Study on the Effect of Terlipressin on Recovery of Liver Function After Hepatectomy: a Multicenter Randomized Controlled Study
Brief Title: The Effect of Terlipressin on Recovery of Liver Function After Hepatectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Terlipressin-Hepatectomy
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Terlipressin Adverse Reaction; Ascites Hepatic; Liver Failure; Acute Kidney Injury
Keywords: hepatectomy; terlipressin; liver failure; acute kidney injury
MeSH Terms: conditions — Liver Failure; Acute Kidney Injury | interventions — Terlipressin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin plus standard care (Experimental): Immediately after hepatectomy, 1 mg terlipressin was given intravenously after hemostasis was achieved. After surgery, participants were routinely managed, and terlipressin were administrated at a dosage of 2 mg per day for 4 days.
  Interventions: Drug: Terlipressin plus standard care
- Standard care (Other): Participants were not administrated with terlipressin during surgery and were routinely managed after surgery.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Terlipressin plus standard care — All the participants received routine care after surgery. Intraoperative 1 mg, and 1 mg q12h from post-operative day 1 through day 4.
  Other Names: terlipressin infusion plus routine care
  Arms: Terlipressin plus standard care
Other: Standard care — All the participants received routine care after surgery only.
  Other Names: routine care
  Arms: Standard care

SUMMARY:
Portal vein hypertension is associated with post-hepatectomy liver failure in patients with liver cirrhosis. Our previous study found that bolus injection of 1 mg terlipressin immediately after hepatectomy decreased portal vein pressure, and post-operative continuous use of terlipressin decreased the amount of abdominal drain. In this multicenter randomized controlled study, we aim to evaluate the effects of terlipressin in the patients who underwent liver resection complicated by portal vein hypertension.

DETAILED DESCRIPTION:
Portal vein hypertension is associated with post-hepatectomy liver failure in patients with liver cirrhosis. Our previous study found that bolus injection of 1 mg terlipressin immediately after hepatectomy decreased portal vein pressure, and post-operative continuous use of terlipressin decreased the amount of abdominal drain. In this multicenter randomized controlled study, we aim to evaluate the effects of terlipressin in the patients who underwent liver resection complicated by portal vein hypertension. The primary outcome is the total abdominal drain on postoperative day (POD) 1 to 3. The secondary outcomes are: (1) the incidence of post-hepatectomy liver failure; (2) post-operative acute kidney injury; (3) the side effects of terlipressin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects signed informed consent.
* An open liver resection is planned.
* Hepatitis B virus infection background.
* Pre-operative liver function is Child-Pugh A.
* Subjects with clinical significance portal vein hypertension or the liver stiffness > 12 kPa before surgery.
* Portal vein pressure > 12 mmHg at 5 min after liver resection.

Exclusion Criteria:

* Age < 18 y or > 75 y.
* Subjects received anti-cancer therapy within 3 months before surgery, or with a history of open or laparoscopic surgery.
* Portal vein tumor thrombus was confirmed by preoperative imaging study.
* Obstruction of biliary tract.
* Pre-operative ALT or AST > 2×ULN.
* A history of myocardial infarction or chronic kidney disease.
* Severe arrhythmia.
* Intraoperative portal vein pressure could not be measured technically.
* Any other contraindications of the terlipressin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The total abdominal drainage | From post-operative day 1 to day 4.
  from postoperative day 1 through day 3.

SECONDARY OUTCOMES:
The incidence of post-hepatectomy liver failure | From post-operative day 1 to day 30.
  based on the criteria of ISGLS 2011.
The incidence of acute kidney injury | From post-operative day 1 to day 30.
  defined as an absolute increase in serum creatinine (Cr) ≥ 0.3 mg/dl (26.5 μmol/L) and/or ≥ 50% from baseline
The side effects of terlipressin | From post-operative day 1 to day 30.
  the incidences of abdominal pain, diarrhea, headache, hyponatremia, and hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Sun, MD&PhD, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Ruijin Hospital Affiliated To Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Eastern Hepatobiliary Surgery Hospital, Second Military Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavallin M, Kamath PS, Merli M, Fasolato S, Toniutto P, Salerno F, Bernardi M, Romanelli RG, Colletta C, Salinas F, Di Giacomo A, Ridola L, Fornasiere E, Caraceni P, Morando F, Piano S, Gatta A, Angeli P; Italian Association for the Study of the Liver Study Group on Hepatorenal Syndrome. Terlipressin plus albumin versus midodrine and octreotide plus albumin in the treatment of hepatorenal syndrome: A randomized trial. Hepatology. 2015 Aug;62(2):567-74. doi: 10.1002/hep.27709. Epub 2015 Feb 13. PMID 25644760
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Background] Chen X, Zhai J, Cai X, Zhang Y, Wei L, Shi L, Wu D, Shen F, Lau WY, Wu M. Severity of portal hypertension and prediction of postoperative liver failure after liver resection in patients with Child-Pugh grade A cirrhosis. Br J Surg. 2012 Dec;99(12):1701-10. doi: 10.1002/bjs.8951. PMID 23132418
- [Background] Saner FH, Canbay A, Gerken G, Broelsch CE. Pharmacology, clinical efficacy and safety of terlipressin in esophageal varices bleeding, septic shock and hepatorenal syndrome. Expert Rev Gastroenterol Hepatol. 2007 Dec;1(2):207-17. doi: 10.1586/17474124.1.2.207. PMID 19072411